CLINICAL TRIAL: NCT04053361
Title: Catheter Ablation of Atrial Fibrillation/Tachycardia in Patients With Pulmonary Hypertension: a Randomised Study
Brief Title: Catheter Ablation of Atrial Fibrillation in Patients With Pulmonary Hypertension Hypertension: a Randomised Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General University Hospital, Prague (Other)
Responsible Party: Principal Investigator, Stepan Havranek, Consultant, General University Hospital, Prague
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GH-18-02-00027-0-202
Record Dates: First submitted 2019-06-28; First posted 2019-08-12 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Pulmonary Hypertension
Keywords: Atrial Fibrillation; Pulmonary Hypertension; Catheter Ablation
MeSH Terms: conditions — Atrial Fibrillation; Hypertension, Pulmonary | interventions — Catheter Ablation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Clinical ablation (Active Comparator): * Cinical arrhythmia is fairly documented AF, pulmonary vein isolation will be performed. If AF persists after this step, electrical cardioversion will be performed.
  * If clinical arrhythmia is fairly documented type 1 AFL, cavo-tricuspid isthmus ablation will be performed.
  * If clinical arrhythmia is AT, it will be induced (if not persistent), identified by means of activation and/or entrainment mapping, and ablated.
  * If clinical arrhythmia is AT that is non-inducible during EP study, no ablation will be done.
  * If other incidental (or induced) AT is observed that can be qualified as non-clinical it will not be targeted unless considered important to ablate at discretion of operator.
  * No induction protocols for other, on top of already ablated, arrhythmias will be attempted.
  Interventions: Procedure: Catheter ablation
- Group B: Clinical plus substrate-based ablation (Experimental): - The initial ablation steps will be identical to those in patients from Group A.
  Supplemental ablation will consist of:
  * Empirical lesion set within right atrium: superior vena cava isolation, posteroseptal bicaval line, and cavo-tricuspid isthmus ablation (if not already ablated)
  AND
  * Homogenization of low-voltage zones (if any) in left / right atrium defined by bipolar voltage <0.5 mV in sinus rhythm or <0.2 mV in AF / AT. The threshold can be adapted in severely diseased atria to delineate reasonably smaller zones (<20% of atrial surface) achievable to ablate.
  * Arrhythmia induction protocol by10-second burst atrial pacing with cycle length of 300 ms decremented by 10 ms up to atrial refractoriness or cycle length of 200 ms.
  * Inducible ATs will be mapped and ablated if feasible. In case of inducible persistent (>5 min) AF, pulmonary vein isolation will be performed if not previously done as per protocol.
  Interventions: Procedure: Catheter ablation

INTERVENTIONS:
Procedure: Catheter ablation — Catheter ablation of atrial fibrillation or atrial tachykardie related to atrial fibrillation with use of radiofrequency energy.

SUMMARY:
Atrial fibrillation (AF) and atrial tachycardia (AT), including type I atrial flutter, are frequently observed in patients with pulmonary hypertension (PH). Catheter ablation of AF / AT has been established as an effective treatment option in selected patients. However, little is known about the efficacy and safety of this approach in patients with PH. It has also been shown that considerable proportion of patients with PH after acutely successful catheter ablation suffer from the recurrence of clinical or newly manifested arrhythmia. We propose a prospective study to compare two ablation strategies in a randomized fashion: radiofrequency catheter ablation targeting only the clinical arrhythmia versus more extensive substrate-based catheter ablation. This project will investigate the clinical outcome of patients with pulmonary hypertension and symptomatic atrial fibrillation / tachycardia who will be randomly allocated to selective versus complex radiofrequency catheter ablation of arrhythmogenic substrate.

ELIGIBILITY:
Inclusion Criteria:

* Pre-capillary PH (PAMP ≥25 mmHg; PAWP ≤15 mmHg) or combined post- a pre-capillary PH (PAMP ≥25 mmHg; PAWP >15 mmHg; DPG ≥7 mmHg and/or PVR >3 W.u.) of any etiology.

Exclusion Criteria:

* Complex congenital heart defects (corrected or uncorrected)
* Isolated post-capillary PH (PAMP ≥25 mmHg; PAWP >15 mmHg; DPG <7 mmHg and/or PVR ≤ 3W.u.)
* Previous catheter ablation for AF / AT / AFL
* Previous or scheduled cardiac surgery-
* NYHA Class IV, cardiogenic shock
* Life expectancy <1 year
* Non-compliance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Arrhythmia recurrence | 3 months
  Documented arrhythmia recurrence >30 s without antiarrhythmic drugs in post-blanking period after the index ablation

SECONDARY OUTCOMES:
On-drugs arrhythmia recurrence | 3 months
  Documented on-drugs arrhythmia recurrence
Symptoms of arrhythmia | 3 months
  Symptoms of arrhythmia by questionare
Change in Quality of life | 6 months
  EQ5D
Mortality | 3 months
  Mortality of any cause
Procedure-related complication rate | 1 day (Once)
  Complications related to catheter ablation
Reablation | 3 months
  Number of repeat catheter ablations if symptoms are ongoing

CONTACTS AND LOCATIONS:
Locations (3):
- Czechia (3):
  - FN Olomouc, Olomouc
  - IKEM, Prague
  - General University Hospital in Prague, Prague

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Havranek S, Fingrova Z, Skala T, Reichenbach A, Dusik M, Jansa P, Ambroz D, Dytrych V, Klimes D, Hutyra M, Kautzner J, Linhart A, Wichterle D. Catheter ablation of atrial fibrillation and atrial tachycardia in patients with pulmonary hypertension: a randomized study. Europace. 2023 May 19;25(5):euad131. doi: 10.1093/europace/euad131. PMID 37178136